CLINICAL TRIAL: NCT06509295
Title: Effect of Calcium Hypochlorite Versus Sodium Hypochlorite as Root Canal Irrigants on Postoperative Pain and Bacterial Reduction in Mandibular Premolars With Necrotic Pulps. A Randomized Clinical Trial.
Brief Title: Effect of Calcium Hypochlorite Versus Sodium Hypochlorite as Root Canal Irrigants on Postoperative Pain and Bacterial Reduction in Mandibular Premolars With Necrotic Pulps. .
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Youmna Yassen, Principle investigator, resident at faculty of dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENDO 3-7-1(10/4/2024)
Record Dates: First submitted 2024-06-24; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Intervention
MeSH Terms: interventions — calcium hypochlorite; Root Canal Irrigants

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calcium Hypochlorite as root canal Irrigant on Postoperative Pain and bacterial load reduction (Placebo Comparator): Treatment with Calcium Hypochlorite as root canal Irrigant
  Interventions: Other: Calcium Hypochlorite as Root Canal Irrigant
- Sodium Hypochlorite as a root Canal Irrigant (Active Comparator): Treatment with Sodium Hypochlorite as root canal Irrigant
  Interventions: Other: Calcium Hypochlorite as Root Canal Irrigant

INTERVENTIONS:
Other: Calcium Hypochlorite as Root Canal Irrigant — Calcium Hypochlorite used as root canal irrigant during chemo-mechanical preparation

SUMMARY:
This study aims to assess the effect of Calcium Hypochlorite Versus Sodium Hypochlorite as Root Canal Irrigants on Postoperative Pain and Bacterial Reduction in Mandibular Premolars with Necrotic Pulps.

ELIGIBILITY:
Inclusion Criteria:

1. Systematically healthy patient (ASA I, II).
2. Age between 20 and 55 years
3. Male or female.
4. Mandibular premolar teeth having single canals diagnosed with pulp necrosis with asymptomatic apical periodontitis.
5. Radiographic examination using Digora intraoral periapical sensor plate and software showing mandibular premolars with (0-2 mm) periapical radiolucency.

Exclusion Criteria:

1. Medically compromised patients having significant systemic disorders. (ASA III or IV).
2. History of intolerance to NSAIDS.
3. Teeth with:

   * Immature roots
   * Vital pulp tissues.
   * Association with swelling.
   * Acute peri-apical abscess or acute exacerbation of a chronic abscess.
   * Mobility Grade II or III.
   * Previously accessed or endodontically treated
   * Deep periodontal pockets more than 4 mm
   * Vertical root fractures, coronal perforation, calcification, and external or internal root resorptions.
4. Patients who could not interpret the NRS.
5. Patients with diabetes, immune-compromising, and immunosuppression disease and pregnant women were, also, excluded.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-29 (Estimated); Primary Completion 2025-04-20 (Estimated); Study Completion 2025-05-29 (Estimated)

PRIMARY OUTCOMES:
Effect of Calcium Hypochlorite Versus Sodium Hypochlorite as Root Canal Irrigants on Postoperative Pain in Mandibular Premolars with Necrotic Pulps. | measured at 6, 12, 24, 48 hours after single visit treatment
  measuring tool: Numerical Rating Scale (NRS). Unite of measurement: Categorical None 0 Mild 1-3 Moderate 4-6 Severe 7-10 Time of measurements: At 6, 12, 24, 48- hours post-treatment.

SECONDARY OUTCOMES:
Effect of Calcium Hypochlorite Versus Sodium Hypochlorite as Root Canal Irrigants on Bacterial Reduction in Mandibular Premolars with Necrotic Pulps. | T0=Baseline immediate after access preparation . T1=Post-instrumentation. T1(within an hour)
  Intracanal bacterial load reduction will be determined by bacterial counting using agar culture technique after root canal preparation (CFUs/ml), The growth will be semi quantitatively determined as very heavy, heavy, moderate, sparse and very sparse depending on the CFU ranging from >100,000,˂100,000,˂10,000,˂1,000, ˂100 colony forming unit per 1 ml BHI respectively.
Number of analgesic tablets taken by the patient after endodontic treatment | Up to 48 hours postoperative.
  Number of analgesic tablets taken by the patient after endodontic treatment Up to 48 hours postoperative.
  Measuring tool: counting Measurment unite: numerical.

IPD SHARING:
Plan to Share IPD: Undecided